CLINICAL TRIAL: NCT02498327
Title: The Efficacy of Red Vine Leaf Extract, Butcher's Broom, Horse Chestnut and Vitamin B6 on the Quality of Life in Females With Chronic Venous Insufficiency
Brief Title: The Efficacy of Venavine Intensive® on the Quality of Life in Females With Chronic Venous Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr, University of Johannesburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: XoliswaRoseMazibuko200729488
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Venous Insufficiency
Keywords: Chronic
MeSH Terms: conditions — Venous Insufficiency; Bronchiolitis Obliterans Syndrome | interventions — Gelatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gelatine Capsules (Placebo Comparator): Gelatine capsules containing only inactive ingredients (starch amyral white, di-calcium phosphate DC and magnesium stearate fine), will be taken once per day, in the morning after breakfast, for 30 days. These capsules will be of identical appearance to the experimental comparator.
  Interventions: Other: Gelatine Capsule
- Venavine Intensive® (Experimental): Gelatine capsules containing the active ingredients of: 360 mg Red Vine Leaf extract, 60 mg of Horse Chestnut extract, 35 mg of Butcher's Broom extract and 3,2 mg of Vitamin B6 as well as the inactive ingredients of starch amyral white, di-calcium phosphate DC and magnesium stearate, will be taken once per day, in the morning after breakfast, for 30 days.
  Interventions: Other: Venavine Intensive®

INTERVENTIONS:
Other: Gelatine Capsule — Gelatine capsules containing only the inactive ingredients of starch amyral white, di-calcium phosphate DC and magnesium stearate fine.
  Arms: Gelatine Capsules
Other: Venavine Intensive® — Gelatine capsules containing 360 mg Red Vine Leaf extract, 60 mg of Horse Chestnut extract, 35 mg of Butchers Broom extract and 3,2 mg of Vitamin B6 as well as the inactive ingredients of starch amyral white, di-calcium phosphate DC and magnesium stearate fine.
  Arms: Venavine Intensive®

SUMMARY:
Chronic Venous Insufficiency (CVI) is impaired venous return which results in lower limbs symptoms that include pain, swelling and dermatologic changes. CVI is a condition that affects both males and females, but is more prevalent in females due to the effect of progesterone on vascular tissue resulting in the dilation of veins. The predisposing factors for CVI include: female gender, long periods of standing, decreased physical activity, obesity, poor nutrition, metabolic syndrome, tight and restrictive clothing as well as advanced age, constipation, pregnancy and ascites. Conventional treatment may involve surgery, compression stockings, laser therapy, sclerotherapy and venoactive drugs, which are aimed at improving the appearance of varicose veins and decreasing pain and swelling.

The combination of Red Vine, Butcher's Broom, Horse Chestnut and Vitamin B6 is an over-the counter herbal preparation, which is used to treat the symptoms associated with CVI. Studies done on each of the preparation's individual constituents demonstrate their efficacy in improving blood circulation, thereby alleviating symptoms associated with venous stasis. The individual extracts improve venous tone and blood circulation, however there are no studies on the combined effect of these individual ingredients and their efficacy on the quality of life of females affected by CVI.

The aim of this study is to determine the efficacy of a combination of Red Vine Leaf extract, Butcher's Broom, Horse Chestnut and Vitamin B6 on the quality of life in female participants with CVI, using the Chronic Venous Insufficiency Quality of Life Questionnaire (CIVIQ-20).

DETAILED DESCRIPTION:
The study is a double-blind, placebo-controlled study of forty female participants, aged thirty to fifty-five years, conducted over a period of ninety days.The research sample will be shared by another Homoeopathy Master's student Fayrooz Karriem who is researching "The efficacy of the combination of Red Vine extract, Butcher's Broom, Horse Chestnut and Vitamin B6 in the treatment of chronic venous insufficiency associated symptoms. Participants will be recruited by means of advertisements at the University of Johannesburg (UJ) Health Clinics.

The research sample will be randomly divided into two groups (X and Y), in matched pairs according to age and severity of symptoms. Participants will select a remedy from one of the boxes, marked with X or Y, thereby allocating themselves to either the experimental group or the control group.

At the first consultation, respondents will undergo a screening test for eligibility to participate in the study. This will be done by means of the inclusion and exclusion criteria. Participants that are eligible to take part in the study will be given an information and consent form to read and sign. If any questions arise, they will be answered by the researcher. A physical examination will be conducted using a modified University of Johannesburg Homoeopathy case taking form. The physical examination will include vital signs and examination procedure for CVI. Participants will be asked to fill in the CIVIQ-20 questionnaire with the assistance of the researcher.

At the end of the first consultation participants will be given either the combination of Red Vine, Butcher's Broom, Horse Chestnut and Vitamin B6 capsules or placebo capsules and will be advised to start taking the capsules the next morning. Participants will be given enough capsules to last them until the next consultation (30 capsules); participants will also be advised not to change their normal routine during the course of the study. If it happens that the participants take aspirin during the course of the study, they will be required to report it to the researcher. Aspirin has anti-coagulant effects which may have an effect on CVI.

On day thirty of the study, participants will have the first follow up consultation. A physical examination will be conducted and participants will fill out the CIVIQ-20 questionnaire based on their experience over the past thirty days. At the end of the first follow up, participants will be given thirty capsules of the herbal combination or placebo (as selected by the participant after the first consultation) to be taken as previously instructed.

On day sixty a second follow up consultation will be conducted and the procedure followed on day thirty will be repeated on day sixty.

The final follow up consultation will be on day ninety, where a physical examination will be conducted and the CIVIQ-20 questionnaire will be completed. On the last day no capsules will be given.

All data collected by the questionnaire, will be statistically analysed with the assistance of a statistician at Statkon, UJ. The between groups comparison will be analysed using the Mann-Whitney U-test. The comparison within the groups will be conducted using the Friedman test and differences over time will be analysed using the Wilcoxon post hoc test.

ELIGIBILITY:
Inclusion Criteria:

* Females between the ages thirty to fifty five years;
* experiencing at least three symptoms from Clinical, Etiology, Anatomy and Pathophysiology (CEAP) Classification C1-C4 of CVI, which includes varicose veins, tired or heavy legs, pain in the legs, tingling calves, venous oedema, induration of the legs, brown discolouration in the legs, skin changes such as erythema in the legs; and
* symptoms must be aggravated by walking/standing and symptoms ameliorated by rest and limb elevation.

Exclusion Criteria:

* Are pregnant or lactating;
* are on chronic medication for cardiovascular disorder;
* have any chronic diseases that are not sufficiently managed;
* are experiencing CEAP C5-C6 of CVI, including venous ulceration;
* are on Warfarin or blood thinning medication;
* have any liver or kidney pathologies;
* are hypersensitive to any/all herbal extracts;
* are on any treatment (herbal or conventional) for CVI; and/or
* are using compression stockings or Kinesio Taping therapy.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The quality of life as measured by the CIVIQ-20 | Every 30 days for 90 days
  The CIVIQ-20 is made up of 20 multiple choice questions subdivided into four categories: psychology, pain, physical repercussion and social repercussions. The questions are equally weighted and the value indicates the degree of deterioration of quality of life; 0 being the highest quality of life and 100 being the lowest. It has been tested to be a reliable measurement tool in evaluating the quality of life in those with CVI.

CONTACTS AND LOCATIONS:
Overall Officials: Radmila Razlog, M.TechHom, Study Director — University of Johannesburg
Locations (1):
- University of Johannesburg, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No